CLINICAL TRIAL: NCT03444064
Title: Polyclonal Regulatory T Cell (PolyTreg) Immunotherapy in Islet Transplantation
Brief Title: PolyTreg Immunotherapy in Islet Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Diabetes Research Institute Foundation (Other); Liana's Dream Foundation (Unknown); Juvenile Diabetes Research Foundation (Other); Alberta Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071320
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
Keywords: Islet transplantation; Diabetes treatment; PolyTregs; Immunotherapy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Participants in this arm receive islet transplant only, and no PolyTregs.
- Treatment (Experimental): Participants in this arm receive PolyTregs infusion at week 6 post islet transplant.
  Interventions: Biological: PolyTregs

INTERVENTIONS:
Biological: PolyTregs — Treatment group receive PolyTregs 6 weeks after islet transplantation as immunotherapy to improve islet survival and reduce the need for immunosuppression drugs.
  Other Names: Ex vivo Expanded Autologous CD4+CD127lo/-CD25+ Polyclonal Regulatory T cells
  Arms: Treatment

SUMMARY:
Islet transplantation is a relatively new procedure used in people with difficult to control Type 1 diabetes. Patients who receive an islet transplant take medication that suppresses their immune system and prevent rejection of the islet tissue. In spite of the strengths of the current immunosuppression regimen, it has failed to enhance single-donor success rates, and the majority of patients require 2 or more islet transplants to achieve insulin independence. The need for life-long, high-dose immunosuppression is also associated with substantial side effects, and continues to limit application of islet transplantation earlier in the course of the disease.

The investigators have learned that Regulatory T cells (Tregs), a small subset of cluster of differentiation 4+ (CD4+) T cells, have emerged as the major contributor to self-tolerance through suppression of activation and effector function of other immune cells. Tregs function by preventing the initiation of unwanted immune activation and by suppressing ongoing immune response to limit bystander tissue destruction. It has been suggested that infusion of Tregs before extensive graft damage may improve long-term graft outcomes.

This study is an open label, controlled, dose finding pilot study. Up to 18 participants will be recruited including 12 participants receiving the investigational treatment and 6 participants being assigned to control group. All participants will undergo the routine Standard of Care islet transplant procedure, and will be maintained on lower dose tacrolimus and sirolimus immunosuppression.

The primary goal is to assess the safety and feasibility of intravenous infusion of ex vivo-selected and ex vivo-expanded autologous PolyTregs in islet transplant patients. The other goal is to assess the effect of Tregs on beta cell function in islet transplant patients.

The control group (6) will receive the current Edmonton islet transplant induction therapy (Alemtuzumab with Etanercept and Anakinra). The intervention group (up to 12) will receive islet transplant with same induction therapy as control group and PolyTregs (400-1600 million) six weeks post- transplant and will be followed for 1 year to assess safety and preliminary efficacy of Treg therapy. The Treg product will be administered via a peripheral intravenous (IV) line primed with saline per established standard operating procedures in approximately 20 to 30 minutes. The intravenous line will be maintained after the infusion and the participant will be asked to remain in the hospital for 24 hours. All participants will be maintained on low dose tacrolimus and sirolimus immunosuppression.

The investigators will also use retrospective data from the islet transplant cohort receiving Tac/mycophenolate mofetil(MMF) with alemtuzumab (>100 patients).

All study participants will be followed up for 58 weeks. Tests and assessments will be performed at each key study visit and will be allowed for +/- 2 weeks to accommodate scheduling.

The following measurements will be recorded at each key study visit :

Blood work, including the following:

Complete blood count (CBC) and differential

Creatinine and electrolytes

Fasting glucose and c-peptide

Any adverse events

Physical examination

Body weight (kg)

Vital signs (BP, HR)

Glucose records for self-monitoring.

Hemoglobin A1c

Insulin use (total daily dose)

Autoantibodies and autoreactive T cell

MMTT

Immune profile

DETAILED DESCRIPTION:
BACKGROUND:

Type 1 diabetes mellitus (T1DM) is an autoimmune disease characterized by the destruction of pancreatic beta (β)-cells, resulting in absolute deficiency of insulin. To date, clinical islet transplantation is an accepted modality to treat select patients who exhibit frequent hypoglycemic events and severe glycemic liability. The "Edmonton Protocol" became a milestone by reporting sustained C-peptide production and high rates of insulin-independence after transplant in patients with T1DM. Due to the challenges associated with allo- and autoimmunity in islet transplantation, appropriate immunosuppression is necessary to prevent acute and/or long-term rejection. Current immunosuppression protocols used in Edmonton and many other international sites for islet transplantation consist of a combination of induction, anti-inflammatory and maintenance therapy, accounting for higher success rates of islet transplantation. In spite of the strengths of the current immunosuppression regimen described above, it has failed to enhance single-donor success rates (15%), with the majority of patients requiring 2 or more islet transplants to achieve insulin independence. In Edmonton, clinical trials are designed to improve islet isolation, engraftment and long-term graft survival. The need for life-long, high-dose immunosuppression is associated with substantial side effects, and continues to limit application of islet transplantation earlier in the course of the disease.

Regulatory T cells (Tregs) are a small subset of CD4+ T cells that depend on the FOXP3 transcription factor for their lineage differentiation and function. Tregs have emerged as the major contributor to self-tolerance through suppression of activation and effector function of other immune cells. Tregs function by preventing the initiation of unwanted immune activation and by suppressing ongoing immune responses to limit bystander tissue destruction. It has been suggested that infusion of Tregs before extensive graft damage may improve long-term graft outcomes. Unlike generalized immunosuppressive regimens, Tregs are long-lived and can function in a dominant and antigen-specific manner. Thus, therapeutic infusion of Tregs has the potential to induce long-term donor-specific tolerance without impeding desired immune responses to pathogens and tumors in transplant patients. In terms of diabetes, both animal and human studies demonstrate the central role of Tregs in preserving β-cell function. Infusion of Tregs prevents and even reverses diabetes in non-obese diabetic (NOD) mice. It has been demonstrated in animal studies that infused Tregs migrate to the allograft site shortly after transplantation and can induce stable islet graft survival without immunosuppression. Recent human studies report functional defects of Tregs in T1DM, which appear to be reversible.

This clinical trial is collaboration between Dr. Shapiro's Clinical Islet Transplantation Program team in Edmonton, Alberta with Drs. Tang and Bluestone's teams at the University of California San Francisco (UCSF). Drs. Tang and Bluestone have been instrumental in developing PolyTreg technology, providing an opportunity for this exciting collaboration in a clinical trial of Treg infusion in islet transplantation. Dr. Tang's team focuses on translating knowledge on mechanisms of immune tolerance into novel therapeutics for treating autoimmune diabetes and preventing transplant rejection. They have demonstrated the efficacy of Tregs at multiple levels to halt tissue destruction in diabetic mouse models by subverting fully differentiated effector T-cells. Dr. Bluestone's research over the past 25 years has focused on understanding the basic processes that control T-cell activation and immune tolerance in autoimmunity and organ transplantation including a special emphasis on Tregs. Dr. Bluestone has demonstrated that PolyTreg immunotherapy can be safely administered in adult patients with new onset T1DM. Drs. Tang and Bluestone have abundant experience in Treg isolation and production and Treg immunotherapy, and bring strong technical and scientific support to this project. The investigators expect that this collaboration will integrate the strengths of both Treg immunotherapy and the standard treatment for islet transplant. Hence, this trial is to investigate the safety and efficacy of Treg infusion incorporated into the current protocol for islet transplantation, in the hope of finding more effective alternatives to the current immunosuppression regimen in islet transplantation.

TRIAL DESIGN

Based on existing pre-clinical and clinical findings, the investigators hypothesize that Tregs protect from both auto and allorejection of transplanted islets, thereby improving insulin independent durability and C-peptide function over time in adults with T1DM.

Primary Objective

To assess the safety and feasibility of intravenous infusion of ex vivo-selected and ex vivo-expanded autologous polyTregs in islet transplant patients.

Primary Outcome Measure/Endpoint

Adverse events

Laboratory abnormalities

Signs of toxicity

Infusion reactions

Complications related to infection

Secondary Objective

To assess effects on endogenous insulin secretion: Assess the effect of Tregs on b cell function in islet transplant patients.

Secondary Outcome Measure/Endpoint

C-peptide response during MMTTs

Insulin use

HbA1C

Exploratory Objective

Surrogate markers of diabetes immune response: Measure the effect of PolyTregs on the pathologic autoimmune and allo-immune responses.

Exploratory Outcome Measure/Endpoint Multicolor flow cytometry (MFC) to assess effect on immune profile (pre- infusion, 1, 2, 4 weeks and 3, 6 and 12 months post-infusion)

Autoantibodies and autoreactive T cell using tetramer/or ELISA spot assay (pre-infusion, and 3, 6 and 12 months post infusion).

Persistence and stability of infused PolyTregs in blood using deuterium labelling (Days 1, 7, 14, 28, 3 months,6 months and 12 months after infusion)

This trial design will allow determination of the following specific aims:

To demonstrate the safety of PolyTreg immunotherapy in islet transplantation in Type 1 diabetic patients.

To assess the immunological impact of PolyTreg immunotherapy on patients receiving islet transplant.

To assess the efficacy and to establish the optimal dose for PolyTreg immunotherapy.

The investigators propose that PolyTregs will protect/dampen both auto and allo-rejection, thereby improving insulin independent durability and C-peptide function over time. In this trial, the investigators propose low level Tac/Sirolimus immunosuppression, the investigators hope that less early exposure and long-term exposure to high dose tacrolimus will lead to marked improvement in Beta cell function, less renal dysfunction, less opportunistic infections, less Posttransplant lymphoproliferative disease (PTLD). The long-term goal is to develop and optimize PolyTreg dosing for a subsequent Phase 2 efficacy/safety randomized controlled trial (RCT).

STUDY PROCEDURES

Study participants will undergo a screening evaluation for this study. This will include the screening for standard of care islet transplant. For women of child bearing potential, the investigators will ask to confirm they are not pregnant with a blood test. If the patient is eligible and has consented to take part, he / she will be assigned into either the control group or treatment group at the investigator's discretion. The only difference between the two groups will be that the treatment group will receive PolyTregs infusion and the control group will not receive PolyTregs infusion. The investigators will collect certain details from his / her medical records, including age, sex, ethnicity and medical information. If the patient is assigned into the treatment group, a blood sample of 400 mL will be collected for PolyTregs manufacturing, which will be infused back to the patient at week 6 after islet transplant. The investigators will enrol two participants in the control group at first and will proceed with further enrolment for both groups if the procedure appears safe in the first two patients.

For treatment group:

Study visit 1: Pre-islet transplant

Before initiation of islet transplant induction therapy, a total of 400 ml whole blood will be collected and immediately transported to the UCSF for PolyTregs manufacturing.

Study visit 2: Islet transplant

At this visit, participants will undergo islet transplant according to the current standard procedures at the University of Alberta Hospital. The only difference will be the use of lower doses of Tacrolimus/Sirolimus for immunosuppression.

Study visit 3: 30 days ± 7 days post-islet transplant

At visit 2, participants will have standard of care metabolic testing and blood samples taken in the Clinical Investigation Unit (CIU) at the University of Alberta Hospital (UAH). These tests assess the function of transplanted islets and include an arginine-stimulated c-peptide test and an Ensure test. Blood samples will be taken at various time intervals over approximately 90 minutes and will test for: HbA1c, c-peptide, insulin and glucose. The investigators may also ask to review participants' insulin usage /blood glucose records. In addition, a blood sample will be collected for the testing of immune profiles, antibodies and T cell function.

Study visit 4: PolyTreg infusion (6 weeks ± 7 days post-islet transplant)

The participant will be admitted to UAH at week 6 post-islet transplantation for PolyTregs infusion. He / she will stay at the UAH for 24 hours for monitoring after the infusion. A blood sample will be collected to assess the persistence and stability of infused PolyTregs while the participant stays in the hospital.

Study visit 5: 1 week ± 2 days post-PolyTregs infusion

A blood sample will be collected at UAH at Day 7 after PolyTregs infusion to assess the persistence and stability of infused PolyTregs and participants' immune profiles.

Study visit 6: 2 weeks ± 4 days post-PolyTregs infusion

A blood sample will be collected at UAH at Day 14 after PolyTregs infusion to assess the persistence and stability of infused PolyTregs and participants' immune profiles.

Study visit 7: 4 weeks ± 7 days post-PolyTregs infusion

A blood sample will be collected at UAH at Day 28 after PolyTregs infusion to assess the persistence and stability of infused PolyTregs and participants' immune profiles.

Study visit 8: 6 weeks ± 7 days post-PolyTregs infusion (12 weeks ± 7 days post-islet transplant)

At this visit, participants will have standard of care metabolic testing and blood samples taken in the CIU at the UAH. These tests assess the function of transplanted islets and include an arginine-stimulated c-peptide test and an Ensure test. Blood samples will be taken at various time intervals over approximately 90 minutes and will test for: HbA1c, c-peptide, insulin and glucose. The investigators may also ask to review participants' insulin usage /blood glucose records.

Study visit 9: 12 weeks ± 7 days post-PolyTregs infusion

A blood sample will be collected at UAH at week 12 after PolyTregs infusion to assess the persistence and stability of infused PolyTregs, immune profiles and antibodies and T cell function.

Study visit 10: 26 weeks ± 30 days post-PolyTregs infusion

A blood sample will be collected at UAH at week 26 after PolyTregs infusion to assess the persistence and stability of infused PolyTregs, immune profiles and antibodies and T cell function.

Study visit 11: 52 weeks ± 30 days post-PolyTregs infusion

A blood sample will be collected at UAH at week 52 after PolyTregs infusion to assess the persistence and stability of infused PolyTregs, immune profiles and antibodies and T cell function. Participants will also have standard of care metabolic testing and blood samples taken in the CIU at UAH. These tests assess the function of transplanted islets and include an arginine-stimulated c-peptide test and an Ensure test. Blood samples will be taken at various time intervals over approximately 90 minutes and will test for: HbA1c, c-peptide, insulin and glucose. The investigators may also ask to review participants' insulin usage /blood glucose records.

Long-term Standard of Care Follow-up

After study visit 11, participants will be followed by the standard of care schedule for islet transplant.

For control group:

Study visit 1: Islet transplant

At this visit, participants will undergo islet transplant according to the current standard procedures at the University of Alberta Hospital. The only difference will be the use of lower doses of Tacrolimus/ Sirolimus for immunosuppression.

Study visit 2: 30 days (± 7 days) post-islet transplant

At visit 2, participants will have standard of care metabolic testing and blood samples taken in the Clinical Investigation Unit (CIU) at the University of Alberta Hospital (UAH). These tests assess the function of transplanted islets and include an arginine-stimulated c-peptide test and an Ensure test. Blood samples will be taken at various time intervals over approximately 90 minutes and will test for: HbA1c, c-peptide, insulin and glucose. The investigators may also ask to review patient's insulin usage /blood glucose records. In addition, a blood sample will be collected for the testing of immune profiles, antibodies and T cell function.

Study visit 3: 7 weeks ± 7 days post-islet transplant

At visit 3, a blood sample will be collected at UAH to assess participants' immune profiles.

Study visit 4: 8 weeks ± 7 days post-islet transplant

At visit 4, a blood sample will be collected at UAH to assess participants' immune profiles.

Study visit 5: 10 weeks ± 7 days post-islet transplant

At visit 5, a blood sample will be collected at UAH to assess participants' immune profiles.

Study visit 6: 12 weeks ± 7 days post-islet transplant

At this visit, participants will have standard of care metabolic testing and blood samples taken in the Clinical Investigation Unit (CIU) at the University of Alberta Hospital (UAH). These tests assess the function of transplanted islets and include an arginine-stimulated c-peptide test and an Ensure test. Blood samples will be taken at various time intervals over approximately 90 minutes and will test for: HbA1c, c-peptide, insulin and glucose. The investigators may also ask to review patient's insulin usage /blood glucose records.

Study visit 7: 18 weeks ± 7 days post-islet transplant

At visit 7, a blood sample will be collected at UAH to assess participants' immune profiles and antibodies and T cell function.

Study visit 8: 32 weeks ± 30 days post-islet transplant

At visit 8, a blood sample will be collected at UAH to assess participants' immune profiles and antibodies and T cell function.

Study visit 9: 58 weeks ± 30 days post-islet transplant

At visit 9, a blood sample will be collected at UAH to assess participants' immune profiles and antibodies and T cell function. Study participants will also have standard of care metabolic testing and blood samples taken in the CIU at UAH. These tests assess the function of transplanted islets and include an arginine-stimulated c-peptide test and an Ensure test. Blood samples will be taken at various time intervals over approximately 90 minutes and will test for: HbA1c, c-peptide, insulin and glucose. The investigators may also ask to review participants' insulin usage /blood glucose records.

Long-term Standard of Care Follow-up

After study visit 9, participants will be followed by the standard of care schedule for islet transplant.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, subjects must be 18-68 years old, and have had T1DM for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

1. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, or a Clarke score ≥4, or HYPO score ≥1000, or lability index (LI) ≥400 or combined HYPO/LI >400/>300.
2. Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.

In addition, participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

Patients will be excluded if they meet any one or more of the following criteria:

1. Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent myocardial infarction (within past 6 months); (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam
2. Active alcohol or substance abuse (must be abstinent for 6 months prior to transplant)
3. Clinical history of T1DM diagnosed >age 40, insulin dependent <5 years
4. Active infection including Hepatitis C, Hepatitis B, HIV, tuberculosis (TB) (subjects with a positive purified protein derivative (PPD) performed within one year of enrolment, and no history of adequate chemoprophylaxis)
5. Measured glomerular filtration rate (GFR) < 60mL/min/1.73 m2
6. Presence or history of macroalbuminuria (>300 mg/g creatinine)
7. Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months)
8. Baseline Hb < 105g/L (<10.5 g/dL) in women, or < 120 g/L (<12 g/dL) in men
9. Untreated proliferative retinopathy
10. Positive pregnancy test, intent for future pregnancy, failure to follow effective contraceptive measures, or presently breast-feeding
11. Previous transplant or evidence of significant sensitization on panel reactive antibody (PRA) (at the discretion of the investigator).
12. Insulin requirement >1.0 U/kg/day
13. HbA1C >12%
14. Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L (133 mg/dL), treated or untreated; and/or fasting triglycerides > 2.3 mmol/L (90 mg/dL)]
15. Under treatment for a medical condition requiring chronic use of steroids
16. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT-INR > 1.5
17. Untreated Celiac disease
18. Patients with a Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 58 weeks
  Any adverse event that occurs during the study

SECONDARY OUTCOMES:
Stimulated C-peptide level | Baseline
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)
Stimulated C-peptide level | Day 30 post islet transplant
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)
Stimulated C-peptide level | Day 90 post islet transplant
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)
Stimulated C-peptide level | Week 58 post islet transplant
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada